CLINICAL TRIAL: NCT02855476
Title: HDClarity: a Multi-site Cerebrospinal Fluid Collection Initiative to Facilitate Therapeutic Development for Huntington's Disease
Acronym: HDClarity
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: CHDI Foundation, Inc. (Other)
Responsible Party: Principal Investigator, Edward Wild, Dr, University College, London
Other Study IDs: 15/0519
Record Dates: First submitted 2016-07-26; First posted 2016-08-04 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF, serum, plasma (participant DNA available via Enroll-HD)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Early Pre-manifest HD: Participants eligible are persons who meet the following criteria:
  1. Are 18-75 years of age, inclusive, at the time of consent; and
  2. Do not have clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score < 4; and
  3. Have CAG expansion ≥ 40; and
  4. Have burden of pathology score, computed as (CAG - 35.5) × age, < 250
- Late Pre-manifest HD: Participants eligible are persons who meet the following criteria:
  1. Are 18-75 years of age, inclusive, at the time of consent; and
  2. Do not have clinical diagnostic motor features of HD, defined as Unified Huntington's Disease Rating Scale (UHDRS) Diagnostic Confidence Score < 4; and
  3. Have CAG expansion ≥ 40; and
  4. Have burden of pathology score, computed as (CAG - 35.5) x age, ≥ 250
- Early Manifest HD: Participants eligible are persons who meet the following criteria:
  1. Are 21-75 years of age, inclusive, at the time of consent; and
  2. Have clinical diagnostic motor features of HD, defined as UHDRS Diagnostic Confidence Score = 4; and
  3. Have CAG expansion ≥ 40; and
  4. Have Stage I or Stage II HD, defined as UHDRS Total Functional Capacity (TFC) scores between 7 and 13 inclusive
- Moderate Manifest HD: Participants eligible are persons who meet the following criteria:
  1. Are 21-75 years of age, inclusive, at the time of consent; and
  2. Have clinical diagnostic motor features of HD, defined as UHDRS Diagnostic Confidence Score = 4; and
  3. Have CAG expansion ≥ 40; and
  4. Have Stage III HD, defined as UHDRS TFC scores between 3 and 6, inclusive
- Advanced Manifest HD: Participants eligible are persons who meet the following criteria:
  1. Are 21-75 years of age, inclusive, at the time of consent; and
  2. Have clinical diagnostic motor features of HD, defined as UHDRS Diagnostic Confidence Score = 4; and
  3. Have CAG expansion ≥ 40; and
  4. Have Stage IV HD, defined as UHDRS TFC scores between 0 and 2, inclusive
- Incomplete Penetrance HD: Participants eligible are persons who meet the following criteria:
  1. Are 18-75 years of age, inclusive, at the time of consent; and
  2. Have CAG expansion of 36-39
- Juvenile Manifest HD: Participants eligible are persons who meet the following criteria:
  1. Are ≥11 years of age at the time of consent; and
  2. Have clinical diagnostic features of juvenile HD, defined as UHDRS Diagnostic Confidence Score = 4 aged ≤20 years; and
  3. Have CAG expansion ≥ 40
- Healthy Control: Participants eligible are persons who meet the following criteria:
  1. Are 18-75 years of age, inclusive, at the time of consent; and
  2. Have no known family history of HD; or
  3. Have known family history of HD but have been tested for the huntingtin gene CAG expansion and are not at genetic risk for HD (CAG < 36).

SUMMARY:
HDClarity will seek at least 2500 research participants at different stages of Huntington's disease (HD). The primary objective is to collect a high quality CSF sample for evaluation of biomarkers and pathways that will enable the development of novel treatments for HD. The secondary objective is to generate a high quality plasma sample collection matching the CSF collections, which will also be used to evaluate biomarkers and pathways of relevance to HD research and development.

DETAILED DESCRIPTION:
This is a longitudinal open-ended observational study. Participants will attend two annual study visits, an Annual Screening Visit followed by an Annual Sampling Visit, and may also attend an optional visit during the first year of enrollment, an Optional Repeat Sampling Visit.

During the Annual Screening Visit, medical history, and clinical and phenotypic data will be obtained. Participants who meet the eligibility requirements of the study and are willing to continue in the study, will return for an Annual Sampling Visit. During that visit, biosamples will be collected following a fast of at least 6 hours, or overnight: blood will be obtained via venipuncture and CSF will be obtained via lumbar puncture. Some participants may be invited to return for an Optional Repeat Sampling Visit approximately 4-8 weeks after the Annual Sampling Visit during their first year of enrolment.

The annual visits are at regular intervals after the first Annual Screening Visit (i.e. at 1, 2, 3 years and so on) ± 2 months. Participants will be encouraged to complete all annual visits; however, they are under no obligation to take part and will be able to skip annual visit without being discontinued from the study. Participants who do not come for an Annual Sampling Visit for three consecutive years will be discontinued from the study, but they may enrol again at a later date, if they so consent. Participants who have already completed HDClarity Sampling Visits under earlier versions of this protocol may also participate in the longitudinal study if they meet the eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-75 years controls, early/late premanifest HD and incomplete penetrance HD, 21-75 years early/moderate/advanced manifest HD, ≥11 years juvenile HD)
* Enroll HD participant
* Capable of consenting or have a legal representative (parent/guardian for juveniles)
* Capable of complying with study procedures
* All participants other than family and community controls must have had a genetic test for HD

Exclusion Criteria:

* Drug trial within 30 days of any sampling visit
* Changes in medication (antidepressant, psychoactive, psychotropic or other medications or nutraceuticals used to treat HD within 30 days)
* Antiplatelet or anticoagulant therapy within 14 days
* Significant comorbidity
* Needle phobia, headache, spinal surgery / deformity
* Clotting or bruising disorder
* Screening blood test abnormalities >10% outside normal range
* Drug / alcohol abuse
* Positive urine pregnancy test at any screening or sampling visit for females of childbearing potential
* Predictable non compliance or unwillingness
* Serious adverse event related to HDClarity study procedures or any lumbar puncture procedure performed for any reason in the previous 30 days

Ages: 11 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants across 8 clinical cohorts will be enrolled at multiple sites up to an estimated minimum of 2500 participants or until the study is terminated by either the Funding Source or Sponsor
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is: | years N/A
  To generate a high quality CSF sample collection for evaluation of biomarkers and pathways that will enable the development of novel treatments for HD.

SECONDARY OUTCOMES:
The secondary objectives of this study are: | years N/A
  To generate a high quality plasma sample collection matching the CSF collections, which will also be used to evaluate biomarkers and pathways of relevance to HD research and development.
  To collect phenotypic and clinical data for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Wild, MA, MB BChir, MRCP, PhD, Principal Investigator — University College, London
Locations (39):
- United States (6):
  - Cenexel, Englewood, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - John Hopkins University, Baltimore, Maryland
  - Wake Forest University, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center, Houston, Texas
- Canada (4):
  - University of British Columbia, The Centre for Huntingtons Disease, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Centre for Movement Disorders, Toronto, Ontario
- France (2):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Le Centre Hospitalier Universitaire de Bordeaux, Bordeaux
- Germany (6):
  - University Hospital Ulm, Ulm, Baden-Wurttemberg
  - Dresden University, Dresden, Saxony
  - St Josef And Elisabeth Hospital, Bochum
  - University Hospital of Erlangen, Erlangen
  - George Huntington Institute, Münster
  - Kbo-Isar-Amper-Klinikum Taufkirchen (Vils), Taufkirchen
- Italy (2):
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan
  - Lega Italiana Ricera Huntington, Rome
- New Zealand (2):
  - The University of Auckland, Grafton, Auckland
  - NZ Brain Research Institute, Christchurch, Canterbury
- Institute of Psychiatry and Neurology, Warsaw, Poland
- Spain (3):
  - Cruces University Hospital, Bilbao, Biscay
  - Hospital de Sant Pau, Barcelona
  - Ramón y Cajal Universitary Hospital, Madrid
- United Kingdom (13):
  - Royal Devon & Exeter NHS Foundation Trust, Exeter, Devon
  - Glasgow Clinical Research Facility, Glasgow, Scotland
  - Birmingham Huntingtons Disease Clinic, Birmingham, West Midlands
  - North Bristol NHS Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff University, Cardiff
  - Fife Health Board - Whyteman's Brae Hospital, Kirkcaldy
  - Leeds Teaching Hospital Trust, Leeds
  - The Walton Centre NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London
  - St George's University Of London, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
The cerebrospinal fluid (CSF) and plasma samples collected in this study will be the basis of future biomarker analysis studies. A Scientific Advisory Committee which will decide how the samples will be analysed.

REFERENCES:
- See also: Study website — http://hdclarity.net
- Available data/document: Study Protocol — http://hdclarity.net/study-information/
- Available data/document: Informed Consent Form — http://hdclarity.net/study-information/ — Draft informed consent form, not yet approved by an Institutional Review Board for clinical use

DOCUMENTS (1):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02855476/Prot_001.pdf